CLINICAL TRIAL: NCT02689362
Title: A Multicenter, Randomized, Double-Blind, Double-Dummy, Active Controlled Clinical Trial for the Validation of Optimum Dose and Preliminary Evaluation of Efficacy and Safety of Evogliptin in Patients With Type 2 Diabetes Mellitus
Brief Title: Evogliptin in Type 2 Diabetes Mellitus (EVOLUTION: EVOgLiptina no Diabetes Mellitus TIpO 2)
Acronym: EVOLUTION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EF144
Record Dates: First submitted 2016-02-10; First posted 2016-02-23 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 4-(3-amino-4-(2,4,5-trifluorophenyl)butanoyl)-3-(tert-butoxymethyl)piperazin-2-one; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Evogliptin 2.5mg+Placebo Sitagliptin (Experimental): Evogliptin (EVO) will be administered orally at a daily dose of: 2.5 mg. The participants randomized to this group will receive 1 tablet daily of EVO 2.5 mg + 1 tablet of sitagliptin (SITA) placebo for 12 weeks.
  Interventions: Drug: Evogliptin; Drug: Placebo Sitagliptin
- Evogliptin 5.0mg+Placebo Sitagliptin (Experimental): Evogliptin (EVO) will be administered orally at a daily dose of: 5.0 mg. The participants randomized to this group will receive 1 tablet daily of EVO 5.0 mg + 1 tablet of sitagliptin (SITA) placebo for 12 weeks.
  Interventions: Drug: Evogliptin; Drug: Placebo Sitagliptin
- Evogliptin 10.0mg+Placebo Sitagliptin (Experimental): Evogliptin (EVO) will be administered orally at a daily dose of: 10.0 mg. The participants randomized to this group will receive 1 tablet daily of EVO 10.0 mg + 1 tablet of sitagliptin (SITA) placebo for 12 weeks.
  Interventions: Drug: Evogliptin; Drug: Placebo Sitagliptin
- Sitagliptin 100mg+Placebo Evogliptin (Active Comparator): SITA at a daily oral dose of 100 mg. The participants randomized to this group will receive 1 tablet daily of SITA 100 mg + 1 tablet of EVO placebo for 12 weeks.
  Interventions: Drug: Sitagliptin; Drug: Placebo Evogliptin

INTERVENTIONS:
Drug: Evogliptin — 1 tablet per day
  Arms: Evogliptin 10.0mg+Placebo Sitagliptin; Evogliptin 2.5mg+Placebo Sitagliptin; Evogliptin 5.0mg+Placebo Sitagliptin
Drug: Sitagliptin — 1 tablet per day
  Arms: Sitagliptin 100mg+Placebo Evogliptin
Drug: Placebo Evogliptin — 1 tablet per day
  Arms: Sitagliptin 100mg+Placebo Evogliptin
Drug: Placebo Sitagliptin — 1 tablet per day
  Arms: Evogliptin 10.0mg+Placebo Sitagliptin; Evogliptin 2.5mg+Placebo Sitagliptin; Evogliptin 5.0mg+Placebo Sitagliptin

SUMMARY:
This phase II, multicenter, randomized, double-blind, double-dummy study with four parallel treatment groups, with active control, will be performed only in brazilian sites under the sponsorship of Eurofarma Laboratórios S.A.. The enrollment for participants in the study will start after the relevant ethical and regulatory approvals and will have an estimated duration of 18 months.

One hundred and forty-four participants with T2DM according to the criteria of ADA who consent to participation in the study by signing the Informed Consent Form (ICF) will be enrolled in the study. In order to be enrolled, the patients must meet all the inclusion criteria and none of the exclusion criteria. The eligible participants will be randomized 1:1:1:1 to receive evogliptin (EVO) at the doses of 2.5 mg/day (N = 36), 5.0 mg/day (N = 36) or 10 mg/day (N = 36) or sitagliptin (SITA) at the dose of 100 mg/day (N = 36), as a single daily dose, for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients meeting all the following criteria will be enrolled in the study:

  1. Aged between 20 and 75 years old.
  2. Diagnosis of T2DM according to the criteria of the American Diabetes Association (ADA).
  3. Not having received treatment with oral hypoglycemic agents or insulin within 12 weeks prior to the screening visit;
  4. Glycated hemoglobin (HbA1c) levels at the screening visit of 7.5% ≤ HbA1c ≤ 10.5%, after appropriate treatment with diet and physical exercise for ≥ 12 weeks;
  5. Body mass index (BMI) of 20 kg/m2 ≤ BMI ≤ 40 kg/m2 at the screening visit.
  6. Signing the Informed Consent Form (ICF) before the performance of any study procedure.

Exclusion Criteria:

- Patients meeting at least one of the following criteria will be excluded from the study:

1. Fasting blood glucose values > 300 mg/dL with severe clinical manifestations present (significant loss weight, severe symptoms and/or ketonuria).
2. Current participation in weight loss programs, with or without anti-obesity drugs use.
3. Presence of heart failure functional class III or IV according to the New York Heart Association (NYHA).
4. Presence of symptomatic liver or gall bladder disease.
5. History of myocardial infarction, transient ischemic attack or coronary angioplasty within 6 months prior to the screening visit.
6. History of gastrointestinal resection.
7. Estimated creatinine clearance (Cockroft and Gault formula) < 60 mL/min.
8. Serum ALT and/or AST level ≥ 2.5 x upper normal limit.
9. Serum CPK level ≥ 3 x upper normal limit.
10. Fasting triglycerides > 400 mg/dL.
11. History of major skin allergy.
12. Use of corticosteroids within 3 months prior to the screening visit.
13. Concomitant treatment with warfarin, dicoumarinic agents or digoxin.
14. Concomitant use of drugs or foods that interfere with the CYP3A4 pathway of liver metabolism including, but not limited to:

    * Inhibitors: antibacterial agents (erythromycin), antifungals (itraconazole, ketoconazole), antivirals (ritonavir, saquinavir, amprenavir, indinavir, nelfinavir), H2 receptor antagonists (cimetidine) and grapefruit juice;
    * Inducers: dexamethasone, rifampin and anticonvulsants (phenytoin, phenobarbital, carbamazepine)
15. History of untreated or uncontrolled thyroid disorder.
16. History of drugs of abuse or moderate/heavy alcohol consumption within 2 months prior to screening.
17. Presence of severe or uncontrolled diseases.
18. Presence of pregnancy or breastfeeding.
19. Women of childbearing potential who do not agree to use a proven effective contraceptive method, unless they are surgically sterile or declare being expressly exempt of pregnancy risk for not engaging in sexual practices or for engaging in them in a non-reproductive manner.
20. Participation in a clinical trial protocol within the previous 12 months unless, at the investigator's discretion, his or her participation may imply a direct benefit for the participant.
21. Presence of any condition which, at the investigator's discretion, may render the patient inadequate for study participation.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-09 (Actual)

PRIMARY OUTCOMES:
Absolute variation of the values obtained in the baseline for the HbA1c | 12 weeks after the start of the treatment

SECONDARY OUTCOMES:
Absolute variation of the values obtained in the baseline for the parameter, fasting blood glucose. | 12 weeks after the start of the treatment
Absolute variation of the values obtained in the baseline for the parameter, body weight. | 12 weeks after the start of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Suely K Inoue, Pharm D, Study Chair — Eurofarma Laboratórios S/A
Locations (10):
- Brazil (10):
  - Centro de Estudos em Diabetes e Hipertensão, Fortaleza, Ceará
  - Hospital Universitário João de Barros Barreto - HUJBB, Belém, Pará
  - CCBR Brasil Centro de Pesquisas e Analises Clinicas Ltda, Rio de Janeiro
  - Centro de Pesquisa Clínica em Diabetes - UNIFESP, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
  - Clinica de Endocrinologia e Metabologia LTDA, São Paulo
  - CPCLIN - Centro de Pesquisas Clinicas LTDA, São Paulo
  - HCFMUSP, São Paulo
  - IMA - Instituto de Pesquisa Clínica e Medicina Avançada Ltda, São Paulo
  - IPEC - Instituto de Pesquisa Clínica Ltda, São Paulo

REFERENCES:
- [Derived] Cercato C, Felicio JS, Russo LAT, Borges JLC, Salles J, Muskat P, Bonansea T, Chacra AR, Eliaschewitz FG, Forti AC. Efficacy and safety of evogliptin in the treatment of type 2 diabetes mellitus in a Brazilian population: a randomized bridging study. Diabetol Metab Syndr. 2019 Dec 19;11:107. doi: 10.1186/s13098-019-0505-z. eCollection 2019. PMID 31890041